CLINICAL TRIAL: NCT05367297
Title: South Asians and Coronary Plaque Registry
Status: Recruiting | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Anand Rohatgi, Professor of Medicine, University of Texas Southwestern Medical Center
Other Study IDs: STU2021-0948
Record Dates: First submitted 2022-04-12; First posted 2022-05-10 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Coronary Artery Disease; Heart Diseases
MeSH Terms: conditions — Coronary Artery Disease; Heart Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Coronary CT Angiogram — A computerized tomography (CT) coronary angiogram is non-invasive imaging test that looks at the arteries that supply blood to your heart.

SUMMARY:
Individuals who self-report as SAs will be recruited to participate in this registry as well as non-SA controls for comparison. All individuals who consent to participate will 1) complete a survey assessing demographics, medical history, family medical history; 2) have blood collection; 3) and CCTA assessment. These data will be combined with clinical data from the electronic health record and, if applicable, the Dallas Hearts and Mind Study and other research studies, for research purposes. The registry will serve to generate primary observations as well as preliminary data for future studies.

DETAILED DESCRIPTION:
To establish a registry of individuals who self-report as South Asian ethnicity with coronary plaque assessment to better understand plaque characteristics in this high-risk group and facilitate future studies investigating the increased coronary disease risk in this population.

South Asian individuals (SAs) are an expanding minority group in the United States (U.S.) with marked excess cardio-metabolic risk. SAs (primarily India, Pakistan, Bangladesh, Nepal, Sri Lanka) are one of the fastest-growing minority groups in the U.S., with an estimated 40% population growth from 2010-2017 (5.4 million in 2017).1-3 SAs in diaspora countries have markedly increased risk of atherosclerotic cardiovascular disease (ASCVD), particularly coronary heart disease (CHD), compared with most other races, ethnicities, and nationalities.4-5 In analysis of census-derived CVD mortality from 2003-2010 across 34 states in the U.S. with over 10 million death records,6 SAs, unlike other Asian groups, had a higher proportionate mortality ratio for ASCVD compared to non-Hispanic White Americans. Similarly, recent data from California revealed an adjusted 2-fold increased incidence of CHD in SA vs. White individuals.7 Moreover, SAs often present with premature ASCVD (7-10 years younger than White persons)8, 9 and more diffuse ASCVD (multiple vascular territories), a consistent finding across diaspora countries.10 The global cardiovascular community has officially recognized SA ethnicity as a "risk-enhancing factor" in the 2018 ACC/AHA Prevention Guidelines11 as well as by incorporating various SA countries of origin in the QRISK2/3 risk calculator used in the U.K.12 Reducing morbidity and mortality from ASCVD in SAs is a clear priority and unmet need.

Prior studies of coronary calcium have not distinguished differences in calcification of coronary artery plaques in this high-risk group, perhaps because arterial plaque calcification is a late-stage process related to aging. Given the premature presentation of coronary disease in SAs and the well-established observation in predominantly White individuals that non-calcified plaque features lead to plaque rupture and myocardial infarction. Therefore, characterizing non-calcified plaque features in SAs may lead to a better understanding of the increased risk in this population and more tailored preventive strategies.

Coronary CT angiogram (CCTA) provide detail information about plaque characteristics and fully assesses both calcified and non-calcified plaque features in the coronary arteries. This information cannot be obtained by any other imaging test and certainly no blood test. CCTA is considered a Class I indication for assessment of chest pain based on its prognostic potential and is a routine test with low risk. The Swedish Cardiopulmonary Bioimage Study used CCTA in 25000 participants without known coronary artery disease to study prevalence, severity and characteristics of coronary atherosclerosis.13 Miami Heart Study, a US based cohort of healthy individuals, performed prospective CCTA measurements in over 2500 participants to understand pathophysiology of subclinical atherosclerosis and investigate its role in genesis of clinical cardiovascular disease.14

Linking novel blood-based markers with these refined plaque features by CCTA may provide a better understanding of what is driving the increased coronary heart disease in South Asians and could lead to earlier prevention and treatment. Since South Asians have a 2-fold higher risk of heart disease and comprise ~60% of all heart disease globally, this is a major clinical problem that deserves increased investigation.

ELIGIBILITY:
Inclusion Criteria:

* Males and Females: Age 18 years or above
* South Asian (SA) adults through self-identification (South Asians to have both biological parents with ancestry from India, Pakistan, Sri Lanka, Nepal and Bangladesh)
* We also propose to enroll an equivalent number of individuals of other descent as a comparator group (Non SA Adult Volunteers)
* Sampling Method: Probability Sample

Exclusion Criteria:

* Under the age of 18 years
* Unable to give informed consent
* Impaired renal function: estimated glomerular filtration rate ≤ 45ml/min
* Baseline heart rate≥70 bpm or ≥66 bpm after beta blocker
* Body mass index (BMI) of 35 or greater
* Prior anaphylactic/non-anaphylactic reaction or other contraindication to iodinated contrast
* Anyone who cannot do CCTA for any reason
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults with South Asian descent (South Asians to have both biological parents with ancestry from India, Pakistan, Sri Lanka, Nepal and Bangladesh) and non South Asian Adult volunteers (age 18 years or older).
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-06-15 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Number and type of adverse and protective CTA-derived plaque features Number and type of adverse and protective CTA-derived plaque features | Day 1
  There will be several features derived from CTA that are validated adverse features, including plaque volume, thin cap, low attenuation, and necrotic core. Protective features include fibrous cap thickness.

CONTACTS AND LOCATIONS:
Overall Officials: Anand Rohatgi, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified demographics, risk factors, clinical history, and research-based measures will be shared with other researchers with appropriate approval.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Data will become available after completed enrollment of any participant. The data will be available for the duration of the registry.
Access Criteria: Researchers may request data from the PI, Dr. Anand Rohatgi. Once approval is given and appropriate regulatory approvals are in place, access may be granted and data shared.